CLINICAL TRIAL: NCT03445130
Title: A Randomized Prospective Placebo-Controlled Study of the Effects of Lavender Aromatherapy on Preoperative Anxiety in Breast Surgery Patients
Brief Title: A Study of the Effects of Lavender Aromatherapy on Preoperative Anxiety in Breast Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-01844
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
Keywords: Preoperative Anxiety; Breast Surgery; Lavender Aromatherapy
MeSH Terms: conditions — Anxiety Disorders | interventions — almond oil; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lavandula Angustifolia oil (LO) (Active Comparator): 2 Drops in Oxygen Mask
  Interventions: Other: Lavandula Angustifolia oil (LO)
- Michelia Alba Leaf oil (MA) (Active Comparator): 2 Drops in Oxygen Mask
  Interventions: Other: Michelia Alba Leaf oil (MA)
- Almond oil (AO) (Active Comparator): 2 Drops in Oxygen Mask
  Interventions: Other: Almond oil (AO)
- Water (Active Comparator): 2 Drops in Oxygen Mask
  Interventions: Other: Water

INTERVENTIONS:
Other: Lavandula Angustifolia oil (LO) — two drops on the inside of an oxygen face mask for 15 minutes.
  Arms: Lavandula Angustifolia oil (LO)
Other: Michelia Alba Leaf oil (MA) — two drops on the inside of an oxygen face mask for 15 minutes.
  Arms: Michelia Alba Leaf oil (MA)
Other: Almond oil (AO) — two drops on the inside of an oxygen face mask for 15 minutes.
  Arms: Almond oil (AO)
Other: Water — two drops on the inside of an oxygen face mask for 15 minutes.
  Arms: Water

SUMMARY:
The purpose of this study is to determine the effects of lavender aromatherapy on preoperative anxiety by measuring changes in pulse rate and anxiety core using Spielberger State-Trait Anxiety Index questionnaires and on postoperative pain medicine usage. Study participants will then be randomized into one of four groups; either they will receive 2 drops of lavender (Lavandula Angustifolia) oil (LO) or 2 drops of Michelia Alba Leaf oil (MA) or 2 drops of unscented Almond oil (AO) or two drops water on the inside of an oxygen face mask for 15 minutes. Linalool makes up ~30% of Lavandula Angustifolia oil and is believed to be its most active anti-anxiety component. Before and after treatment, anxiety level will be measured using the Spielberger State-Trait Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Women, older than 18, American Society of Anesthesiologists (ASA) classification I-III, undergoing elective breast surgery on Tisch 10th floor Day Surgery. Cancer patients are included.

Exclusion Criteria:

* History of asthma, bronchitis, COPD, contact dermatitis to cosmetic fragrances, positive patch test, pregnancy, and significant laboratory abnormalities.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing breast surgery
Enrollment: 200 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Reduction in anxiety as measured by the change in baseline STAI scores | 20 Minutes
  Spielberger State-Trait Anxiety Inventory (STAI) is a self-reported instrument. It was designed to assess levels of state anxiety and traint anxiety, through 40 items scored by a likert-scale. State anxiety can be defined as a transient momentary emotional status that results from situational stress.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wajda, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification. Researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Requests should be directed to Lola.Franco@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.